CLINICAL TRIAL: NCT01940029
Title: Pharmacokinetic Study in Neurosurgical ICU Patients -Using Vancomycin as an Example
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201105079RC
Record Dates: First submitted 2013-08-21; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Neurosurgery, Critical Ill
Keywords: vancomycin, neurosurgery, critical ill, pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, Cerebrospinal fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
Neurosurgical ICU patients often receive hyperosmotic diuretics or cerebrospinal fluid (CSF) drainage to decrease their intracranial pressure. It is also common to keep them under normovolemia or mild hypervolemia status for stable cerebral perfusion pressure (CPP). These patients have large urine output on average, and can decrease the reabsorption of specific medicines by renal tubules. Besides, hypervolemia status might increase the volume of distribution for hydrophilic medicines, and lower their serum concentration. Therefore, the pharmacokinetic characteristics in this population may be different from general population, which impacts the efficacy and toxicity of medicines with narrow therapeutic index.

Vancomycin is used mainly for MRSA (methicillin-resistant S. aureus) infection, and possesses a significant place of therapy in treatment of neurosurgical patients' post-operation infection. The serum concentration of vancomycin exhibits a clear relevance to its efficacy and toxicity. From the investigators' preliminary research of the disposition of vancomycin in neurosurgical ICU patients, the investigators found that their vancomycin serum concentrations were lower than expected, which can be attributed to their 40% higher mean vancomycin clearances than that of neurosurgical general ward patients. However, no definite mechanism leading to this phenomenon was confirmed.

In this study, the investigators prospectively recruit a cohort of adult neurosurgical ICU patients to validate the investigators' preliminary pharmacokinetic parameter models for vancomycin. Furthermore, the investigators will also demonstrate the contribution of different vancomycin elimination routes, renal and CSF drainage eliminating routs, to its total clearance, and the relationship between vancomycin renal clearance and creatinine clearance. Exclusion criteria include renal failure, unstable renal function, obesity, shock status, third space fluid accumulation, burn and pregnancy. The models to validate are used for empirical vancomycin dosage calculation. Therapeutic drug monitoring (TDM) is conducted after vancomycin serum concentration achieves steady state, and the predicted and observed serum concentration of vancomycin are compared to evaluate the consistency. On the other hand, vancomycin excreted from urine and CSF drainage fluid would be calculated to see their independent contribution for total vancomycin clearance. Meanwhile, the investigators try to investigate the mechanism for renal elimination of vancomycin by its association to creatinine clearance values calculated from urine creatinine concentration data.

Bringing all the information together, the investigators hope to provide helpful information for the clinical pharmacokinetics of vancomycin therapy in neurosurgical patients, and to optimize empirical vancomycin dosing and improve treatment success. Through this study, the investigators also wish to understand the possible pharmacokinetic change of other medicines in this population, and provide an important source of reference for clinical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgical ICU patients((therapeutic dose monitoring, TDM))

Exclusion Criteria:

* Non-Neurosurgical ICU patients,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgical ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Vancomycin clearance (Cl) and volume of distribution (Vd) | peak level is drawn at 2 hours post infusion, trough level is drawn before the next dose
  Observed pharamcokinetic parameters will be compared to model predicted pharmacokinetic parameters, to analyze the accuracy and precision of the pharmacokinetic models derived in preliminary studies.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Li Jiuan, Ph.D, Study Chair — Department of Pharmacy, National Taiwan University Hospital